CLINICAL TRIAL: NCT05694754
Title: Transcranial Magnetic Stimulation and Its Effects on Mayor Depressive Disorder and Smoking Cessation
Brief Title: Transcranial Magnetic Stimulation Theta Burst (TMS), Depression and Smoking.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Julian Reyes López (Other)
Responsible Party: Sponsor-Investigator, Dr. Julian Reyes López, Professor, Universidad Autonoma de Queretaro
Organization: Universidad Autonoma de Queretaro (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-03-2022
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder; Smoking Reduction
Keywords: Transcranial magnetic stimulation; Theta Burst; Depression; Tobacco; suicide ideation
MeSH Terms: conditions — Depressive Disorder, Major; Smoking Reduction; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 session (Experimental): Participants will receive 1 session from monday to friday,during 4 weeks, with 600 total pulses per session
  Interventions: Device: Theta Burst Transcranial Magnetic Stimulation
- 3 sessions (Experimental): Participants will receive 3 sessions from monday to friday,during 4 weeks, with 1800 total pulses per session with a 10 minutes rest interval
  Interventions: Device: Theta Burst Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Theta Burst Transcranial Magnetic Stimulation — Magventure MagPro R30 stimulation Device, MCF-B70 stimulation Coill

SUMMARY:
This study evaluates de efficacy of Theta Burst Transcranial Magnetic Stimulation (TMS) applied on the left dorsolateral prefrontal cortex in patients with Major Depressive disorder and tobacco consumption.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) affects 350 million worldwide causing damage on quality of life and risk behavior such as suicide and smoking. smoking is the second leading cause of death causing about 5 million deaths annually. Theta Burst Stimulation (TBS) is a more tolerable protocol administered at lower intensities and shorter intervals than conventional rTMS protocols.

ELIGIBILITY:
Inclusion Criteria:

* With dependence on tobacco use, with depressive symptomatology, that they agree to sign the informed consent letter.

Exclusion Criteria:

* History of head trauma with loss of consciousness, with intracranial metallic objects or metallic plates in the skull, patients with structured suicidal ideation or recent attempts, who suffer from uncontrolled chronic diseases at the time of entering the study (for example: hypertension, diabetes, rheumatic diseases), patients with psychotic symptoms. subjects with alterations in electroencephalogram (epileptiform activity), patients with any type of uncontrolled chronic medical or neurological disease, pregnant women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
MINI Neuropsychiatric Interview | 15 minutes
  It is a short structured diagnostic interview that explores the main psychiatric disorders of Axis I of DSM-IV and ICD-10
Fagerström test | 5 minutes
  it is a short and simple test consisting of 6 questions. The score ranges from 0-10, so that the higher the score, the greater the dependency. Not only does this test measure physical dependence but it also has therapeutic and prognostic value.
Richmond Test | 5 minutes
  Scale consisting of 4 items to assess the degree of motivation to quit smoking on a scale of 1 to 10. For an individual to have expectations of success in a smoking cessation program, they must present a score of 9 or 10 points
Glover-Nilsson Test | 8 minutes
  Test consisting of 11 items to measure the psychosocial and behavioral dependence of individuals; it is scored from 0 to 4, with 4 being the maximum score, items 1,4 and 5 measure psychological dependence, questions 2,3,6,7,8,9 and 10 measure behavioral dependence and question 11 measures social dependence.
Test of the Unit of the Institute of Public Health of Madrid (UISPM) | 10 minutes
  Test consisting of 23 items divided into 6 modules (stimulation, sedation, automatism, social dependency, psychic dependency and gestural dependency) each item is scored from 0 to 4 being 4 the highest score.
Minnesota Nicotine Withdrawal Syndrome Scale (MNWS) | 5 minutes
  This eight-item scale measures withdrawal symptoms (craving, irritability, anxiety, difficulty concentrating, restlessness, increased appetite or weight gain, depression, and insomnia), The score ranges from 0 to 4, with 4 being the highest score, indicating a severe withdrawal syndrome
Nicotine Craving Questionnaire (CCN) | 8 minutes
  12-item questionnaire to assess the degree of craving, with five response options ranging from completely disagree 1 to completely agree 5
Paradigm of reactivity to signals and heart rate variability | 10 minutes
  it consists of presenting a series of images that were chosen from the International Series of images for smoking (with neutral counterparts), Version 1.2 (58), the images were presented as follows : 2 blocks of smoking images and 2 blocks with neutral images that are interspersed, each block contains 25 images with a duration of 6 seconds per image, the test has a total duration of 10 minutes; while the participant observes the images, they will place a polar model H10 bluetooh chest strap sensor to measure HRV
Co-oximetry | 1 minute
  spectrophotometric technique to detect the loss in the oxygenation capacity of hemoglobin that consists of determining the level of carbon monoxide (CO) in the air exhaled by an individual, levels of 10 or more ppm of CO in the exhaled air correspond to smoking subjects. Levels of 6 to 10 ppm in sporadic smokers, and figures below 6 ppm in non-smokers.
Hamilton Rating Depression Scale (HDRS) | 10 minutes
  21 item, Clinical assessment of depressive symptoms
Montgomery-Asberg Rating Depression Scale (MADRS) | 10 minutes
  10 ítem Clinical assessment of the principal depressive symptoms
Hamilton Anxiety Rating Scale (HARS) | 10 minutes
  14 Ítem clinical scale for rating anxiety symptoms.
Beck Depression Invetory (BDI) | 10 minutes
  it´s a 21 ítem self evaluated symptomatology of depression
Beck Hopelesness Scale (BHS) | 10 minutes
  is a 20-item self-report inventory designed to measure 3 major aspects of hopelessness (Feelings about the future, loss of self-motivation and expectations)
Plutchik Risk Suicide Scale | 10 minutes
  it´s a 26 ítem self-reported scale that assess the intensity of suicidal ideation
Beck suicidal ideation scale (BSIS) | 10 minutes
  is an evaluation of suicidal thinking: is an evaluation of suicidal thinking that helps identify individuals at risk of comitting self harm
Wisconsin Card Sorting Test (WCST) | 20 minutes
  is a neuropsychological test that assess cognitive flexibility
Stop Signal Task | 25 minutes
  is a unique versión of a classic approach to measuring response inhibition

SECONDARY OUTCOMES:
Marlowe and Crowne Social Desirability Scale | 10 minutes
  self-applied scale consisting of 33 items for the evaluation of the need for social approval, for example, generating a good impression through socially appropriate responses

CONTACTS AND LOCATIONS:
Overall Officials: Julian V. Reyes López, PhD, Study Director — Universidad Autónoma de Querétaro
Locations (1):
- Sofia Cañizares Gómez, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fluharty M, Taylor AE, Grabski M, Munafo MR. The Association of Cigarette Smoking With Depression and Anxiety: A Systematic Review. Nicotine Tob Res. 2017 Jan;19(1):3-13. doi: 10.1093/ntr/ntw140. Epub 2016 May 19. PMID 27199385
- [Result] Picciotto MR, Mineur YS. Molecules and circuits involved in nicotine addiction: The many faces of smoking. Neuropharmacology. 2014 Jan;76 Pt B(0 0):545-53. doi: 10.1016/j.neuropharm.2013.04.028. Epub 2013 Apr 28. PMID 23632083
- [Result] Ahern E, Kinsella S, Semkovska M. Clinical efficacy and economic evaluation of online cognitive behavioral therapy for major depressive disorder: a systematic review and meta-analysis. Expert Rev Pharmacoecon Outcomes Res. 2018 Feb;18(1):25-41. doi: 10.1080/14737167.2018.1407245. Epub 2017 Nov 30. PMID 29145746
- [Result] Garcia-Gomez L, Hernandez-Perez A, Noe-Diaz V, Riesco-Miranda JA, Jimenez-Ruiz C. SMOKING CESSATION TREATMENTS: CURRENT PSYCHOLOGICAL AND PHARMACOLOGICAL OPTIONS. Rev Invest Clin. 2019;71(1):7-16. doi: 10.24875/RIC.18002629. PMID 30810545
- [Result] Baeken C, Marinazzo D, Everaert H, Wu GR, Van Hove C, Audenaert K, Goethals I, De Vos F, Peremans K, De Raedt R. The Impact of Accelerated HF-rTMS on the Subgenual Anterior Cingulate Cortex in Refractory Unipolar Major Depression: Insights From 18FDG PET Brain Imaging. Brain Stimul. 2015 Jul-Aug;8(4):808-15. doi: 10.1016/j.brs.2015.01.415. Epub 2015 Feb 7. PMID 25744500
- [Result] Arikan MK, Gunver MG, Tarhan N, Metin B. High-Gamma: A biological marker for suicide attempt in patients with depression. J Affect Disord. 2019 Jul 1;254:1-6. doi: 10.1016/j.jad.2019.05.007. Epub 2019 May 6. PMID 31082626
- [Result] Mahoney JJ 3rd, Hanlon CA, Marshalek PJ, Rezai AR, Krinke L. Transcranial magnetic stimulation, deep brain stimulation, and other forms of neuromodulation for substance use disorders: Review of modalities and implications for treatment. J Neurol Sci. 2020 Nov 15;418:117149. doi: 10.1016/j.jns.2020.117149. Epub 2020 Sep 20. PMID 33002757
- [Result] Filipcic I, Milovac Z, Sucic S, Gajsak T, Filipcic IS, Ivezic E, Aljinovic V, Orgulan I, Penic SZ, Bajic Z. Efficacy, Safety and Tolerability of Augmentative rTMS in Treatment of Major Depressive Disorder (MDD): A Prospective Cohort Study in Croatia. Psychiatr Danub. 2017 Mar;29(1):31-38. doi: 10.24869/psyd.2017.31. PMID 28291972
- [Result] Czeisler ME, Lane RI, Petrosky E, Wiley JF, Christensen A, Njai R, Weaver MD, Robbins R, Facer-Childs ER, Barger LK, Czeisler CA, Howard ME, Rajaratnam SMW. Mental Health, Substance Use, and Suicidal Ideation During the COVID-19 Pandemic - United States, June 24-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 14;69(32):1049-1057. doi: 10.15585/mmwr.mm6932a1. PMID 32790653